CLINICAL TRIAL: NCT00556478
Title: A Phase IIb, Multi-center, Randomized, Double-blind, Placebo-controlled Study, With Open-label Follow on, to Evaluate the Efficacy, Safety and Tolerability of PSD502 in Subjects With Premature Ejaculation (PE)
Brief Title: Efficacy, Safety and Tolerability of PSD502 (a Topical Anesthetic) in the Treatment Premature Ejaculation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Plethora Solutions Ltd (Industry)
Collaborators: Shionogi Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSD502-PE-002
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Premature Ejaculation
Keywords: Premature Ejaculation; Lidocaine; Prilocaine; EMLA® cream; topical anesthetics
MeSH Terms: conditions — Premature Ejaculation | interventions — Lidocaine, Prilocaine Drug Combination; Prilocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Double-Blind Active (Active Comparator): Double-blind Phase: Subjects will be randomised to PSD502 respectively if the patient meets all the entry criteria.
  Interventions: Drug: PSD502, contains a mixture of lidocaine and prilocaine
- Double-Blind Placebo (Placebo Comparator): Double-blind Phase: Subjects will be randomised to Placebo respectively if the patient meets all the entry criteria.
  Interventions: Drug: Placebo
- Open Label Phase (Active Comparator): Subjects will all receive PSD502 if they wish to continue in the trial.
  Interventions: Drug: PSD502, contains a mixture of lidocaine and prilocaine

INTERVENTIONS:
Drug: PSD502, contains a mixture of lidocaine and prilocaine — PSD502 spray contains a mixture of lidocaine and prilocaine with Norflurane (HFA-134a) is used as both propellant and solvent. A single dose consists of 3 sprays applied to the glans penis.
  Approximately 5 minutes before intercourse the study spray can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
  Arms: Double-Blind Active; Open Label Phase
Drug: Placebo — The placebo is a metered dose aerosol spray that is identical in appearance to the active treatment and contains the same propellant (norflurane) but has no lidocaine or prilocaine.
  Approximately 5 minutes before intercourse the study spray can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing.
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
  Arms: Double-Blind Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and tolerability of the investigational drug, PSD502 in subjects with premature ejaculation (PE) The study drug, PSD02, is a metered dose (measured dose), topical (applied to the skin surface) anesthetic (numbing) spray containing a mixture of lidocaine and prilocaine. The study drug will be applied in a spray to the penis prior to intercourse in order to decrease sensitivity in an attempt to delay ejaculation.

DETAILED DESCRIPTION:
Most studies evaluating treatments PE include intravaginal ejaculatory latency time (IELT) in the definition of PE. It has been estimated that PE affects 30-40% of the male population, but is paradoxically a condition for which they are least likely to seek help.

Men with PE exhibit abnormal autonomic reflex pathways for the ejaculatory process. These include lower vibratory threshold to ejaculation, shorter bulbocavernous latency time and higher bulbocavernous evoked potentials. Reducing the heightened sensitivity of the glans penis with topical anesthetics might therefore be a way of improving IELT, without adversely affecting the sensation of ejaculation.

Although IELT is an objective measure of ejaculatory function it does not address the impact of therapy on patients' well being and confidence in their sexual performance, which are important markers of treatment benefit. Therefore, if IELT is used as a sole efficacy measure it may not fully characterise the treatment benefit to the patient. For this reason, a patient reported outcome (PRO) known as the Index of Premature Ejaculation (IPE) will be used in this study in conjunction with IELT to evaluate efficacy. Thus the combination of the objective measure of ejaculatory latency with the PRO of IPE should be able to provide efficacy data which are representative of clinical benefit to the patient.

The use of lidocaine, prilocaine and EMLA® cream as topical anesthetics is well established. Many years of experience of use in large numbers of patients, as well as comprehensive non-clinical safety testing programs for various formulations of lidocaine and prilocaine exist, to support their safety and tolerability. This information, together with the clinical data from 3 studies with PSD502 (ANAE-059-00, PSD502-PE-001, and PSD502-PE-003), suggest that PSD502 may have beneficial effects in reducing penile sensation and prolonging IELT, and its use is unlikely to be associated with significant clinical safety or tolerability concerns.

The aim of this study is to provide additional placebo-controlled efficacy data to establish the clinical utility of PSD502 in the treatment of PE. In addition, long term open-label efficacy and safety data will be collected, to further support the registration package for PSD502 in the indication of treatment of PE.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Male and aged 18 years and over.
* Diagnosed with PE according to DMS-IV criteria and ISSM definition
* Diagnosed with lifelong PE
* Acceptable response to Baseline PEP
* Subject must be in a stable heterosexual and monogamous relationship and the partner must provide consent
* Acceptable sexual encounters in the Baseline period.

Exclusion Criteria:

* Subject, or his sexual partner, has received an investigational (non-registered) drug within 30 days of Screening.
* Subject has erectile dysfunction
* The subject, or his sexual partner, has a physical or psychological condition that would prevent them from undertaking the study procedures, including, but not limited to, the following:

  * Urological disease
  * Ongoing significant psychiatric disorder not controlled by medication.
* Subject has safety testing abnormalities at the Screening Visit
* Subjects taking excluded medications or receiving any treatment for PE
* Subject, or his sexual partner, has a current history of alcohol or drug abuse,
* The subject, or his sexual partner, is unlikely to understand or be able to comply with study procedures, for whatever reasons.
* Subject, or his sexual partner, has known drug sensitivity to amide-type local anesthetics.
* Subjects with pregnant partners
* Subject with sexual partners of child-bearing potential and not using appropriate contraception
* Subject, or his sexual partner, has a history of Glucose-6-Phosphate Dehydrogenase (G-6-PD) deficiency or use of medications that would increase susceptibility to methemoglobinemia (e.g. anti-malarial agents).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Culley Carson, MD, Principal Investigator — University of North Carolina
Locations (1):
- Department of Urology, University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinsmore WW, Hackett G, Goldmeier D, Waldinger M, Dean J, Wright P, Callander M, Wylie K, Novak C, Keywood C, Heath P, Wyllie M. Topical eutectic mixture for premature ejaculation (TEMPE): a novel aerosol-delivery form of lidocaine-prilocaine for treating premature ejaculation. BJU Int. 2007 Feb;99(2):369-75. doi: 10.1111/j.1464-410X.2006.06583.x. Epub 2006 Nov 24. PMID 17129234
- [Background] Morales A, Barada J, Wyllie MG. A review of the current status of topical treatments for premature ejaculation. BJU Int. 2007 Sep;100(3):493-501. doi: 10.1111/j.1464-410X.2007.07051.x. Epub 2007 Jul 3. PMID 17608824
- [Background] Henry R, Morales A. Topical lidocaine-prilocaine spray for the treatment of premature ejaculation: a proof of concept study. Int J Impot Res. 2003 Aug;15(4):277-81. doi: 10.1038/sj.ijir.3901011. PMID 12934056

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-Blind Active / Open-Label Active: Double-blind Phase: Subjects will be randomised in a 2:1 ratio of PSD502 or placebo respectively if the patient meets all the entry criteria.
  PSD502, contains a mixture of lidocaine and prilocaine: PSD502 spray contains a mixture of lidocaine and prilocaine with Norflurane (HFA-134a) is used as both propellant and solvent. A single dose consists of 3 sprays applied to the glans penis.
  Approximately 5 minutes before intercourse the study spray (PSD502 or Placebo) can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
- Double-Blind Placebo / Open-Label Active: Double-blind Phase: Subjects will be randomised in a 2:1 ratio of PSD502 or placebo respectively if the patient meets all the entry criteria.
  PSD502 Placebo: The placebo is a metered dose aerosol spray that is identical in appearance to the PSD502 spray and contains the same propellant (norflurane) but has no lidocaine or prilocaine.
  Approximately 5 minutes before intercourse the study spray (PSD502 or Placebo) can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing.
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
Period: Double-blind Phase
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Started | 171 | 85
ITT | 167 | 82
Completed | 150 | 77
Not Completed | 21 | 8
Period: Open-Label Phase
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Started | 146 | 77
Treated in Open-label | 142 | 71
Completed | 132 | 67
Not Completed | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active | Total
Number analyzed (Participants) | 167 | 82 | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 163 | 81 | 244
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.71) | 37.9 (11.97) | 38.7 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 167 | 82 | 249
Region of Enrollment [Number; unit: participants]
  Poland | 68 | 32 | 100
  Canada | 14 | 7 | 21
  United States | 85 | 43 | 128

OUTCOME MEASURES:

1. Primary Outcome: Mean Intravaginal Ejaculatory Latency Time (IELT): Change From Baseline to During 3 Month Double Blind-treatment
Description: To evaluate efficacy of treatment with PSD502 compared with placebo in subjects with PE as measured by:
  • change in mean IELT from baseline to during the 3 month double-blind treatment
  Results provide are ratio (over the 3 months/baseline).
Time Frame: Baseline to 3 Months
Population: ITT
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
ratio | 4.607 [0.01 to 559.78] | 1.505 [0.27 to 12.58]
Statistical Analysis 1: Comparison: Double-Blind Active / Open-Label Active vs Double-Blind Placebo / Open-Label Active; Test type: Superiority or Other; p < 0.0001, ANCOVA; Ratio (over 3 months/Baseline) = 3.05, 95% CI 2-sided [2.29 to 4.06]

2. Primary Outcome: Index of Premature Ejaculation (IPE): Change From Baseline to End of Month 3
Description: To Evaluate Efficacy of Treatment With PSD502 Compared With Placebo in Subjects With PE as measured by:
  • changes in all 3 IPE domains from baseline to month 3
  Ejaculatory control scores range from 4 to 20 with a higher score indicating greater ejaculatory control Sexual satisfaction scores range from 4 to 20 with a higher score indicating greater sexual satisfaction Distress scores range from 2 to 10 with a higher score indicating less distress
Time Frame: Baseline to 3 Months
Population: ITT
Measure: Mean (Full Range); unit: Score
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
Score
  Ejaculatory control | 7.2 [-3 to 16] | 2.2 [-1 to 14]
  Sexual satisfaction | 6.6 [-8 to 16] | 2.1 [-4 to 14]
  Distress | 3.5 [-2 to 8] | 0.9 [-2 to 6]
Statistical Analysis 1: Comparison: Double-Blind Active / Open-Label Active vs Double-Blind Placebo / Open-Label Active; Analysis of IPE domain ejaculatory control; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 5, 95% CI 2-sided [3.61 to 6.34]
Statistical Analysis 2: Comparison: Double-Blind Active / Open-Label Active vs Double-Blind Placebo / Open-Label Active; IPE domain sexual satisfaction; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [3.30 to 5.84]
Statistical Analysis 3: Comparison: Double-Blind Active / Open-Label Active vs Double-Blind Placebo / Open-Label Active; IPE domain distress; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [1.86 to 3.20]

3. Secondary Outcome: Percentage of Subjects With Mean Intravaginal Ejaculatory Latency Time (IELT) > 1 Minute and >2 Minutes During the 3 Months of Double-blind Treatment
Description: Percentage of subjects with mean IELT > 1 minute and >2 minutes during the 3 months of double-blind treatment as measured by the proportion of subjects
Time Frame: 3 months
Population: ITT
Measure: Number; unit: percentage of subjects
Groups:
- Double-Blind Active / Open-Label Active: Double-blind Phase: Subjects will be randomised to PSD502 respectively if the patient meets all the entry criteria.
  PSD502, contains a mixture of lidocaine and prilocaine: PSD502 spray contains a mixture of lidocaine and prilocaine with Norflurane (HFA-134a) is used as both propellant and solvent. A single dose consists of 3 sprays applied to the glans penis.
  Approximately 5 minutes before intercourse the study spray can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
- Double-Blind Placebo / Open-Label Active: Double-blind Phase: Subjects will be randomised to Placebo respectively if the patient meets all the entry criteria.
  Placebo: The placebo is a metered dose aerosol spray that is identical in appearance to the active treatment and contains the same propellant (norflurane) but has no lidocaine or prilocaine.
  Approximately 5 minutes before intercourse the study spray can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing.
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
percentage of subjects
  IELT > 1 minute | 80.2 | 37.8
  IELT > 2 minutes | 57.5 | 14.6

4. Secondary Outcome: Change in Mean Intravaginal Ejaculatory Latency Time (IELT) From Baseline to Month 3
Description: Summary of mean IELT at Baseline and at month 3 during double-blind treatment
Time Frame: 3 months
Population: ITT
Measure: Geometric Mean (Standard Deviation); unit: Seconds
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
Seconds | 140.964 (463.97) | 49.615 (91.75)

5. Secondary Outcome: Change in the Index of Premature Ejaculation (IPE) Domains of Ejaculatory Control, Distress and Sexual Satisfaction From Baseline to Month 1
Description: Change in the IPE domains of ejaculatory control, distress and sexual satisfaction from Baseline to month 1.
  Ejaculatory control scores range from 4 to 20 with a higher score indicating greater ejaculatory control Sexual satisfaction scores range from 4 to 20 with a higher score indicating greater sexual satisfaction Distress scores range from 2 to 10 with a higher score indicating less distress
Time Frame: 1 month
Population: ITT
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
Score
  Ejaculatory control | 5.7 (5.92) | 1.3 (2.75)
  Distress | 2.5 (2.64) | 0.6 (1.70)
  Sexual satisfaction | 5.1 (5.86) | 1.8 (3.54)

6. Secondary Outcome: Subject PEP at Month 1
Description: Scores for perceived control over ejaculation, personal distress related to ejaculation, satisfaction with sexual intercourse and interpersonal difficulty related to ejaculation based on the subject PEP at month 1. Percentage of subjects with at least a 1 point category improvement in subject PEP domain scores at month 1.
Time Frame: 1 month
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
percentage of participants
  Control | 59.6 | 23.5
  Distress | 63.4 | 27.2
  Sexual satisfaction | 62.7 | 33.3
  Interpersonal difficulty | 72.0 | 51.9

7. Secondary Outcome: Change in the Index of Premature Ejaculation (IPE) Domains of Ejaculatory Control, Distress and Sexual Satisfaction From Baseline to Month 2
Description: Change in the IPE domains of ejaculatory control, distress and sexual satisfaction from Baseline to month 2
  Ejaculatory control scores range from 4 to 20 with a higher score indicating greater ejaculatory control Sexual satisfaction scores range from 4 to 20 with a higher score indicating greater sexual satisfaction Distress scores range from 2 to 10 with a higher score indicating less distress
Time Frame: 2 months
Population: ITT
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
Score
  Control | 6.5 (6.06) | 1.4 (3.12)
  Satisfaction | 5.8 (6.19) | 1.3 (3.68)
  Distress | 2.9 (3.00) | 0.7 (1.85)

8. Secondary Outcome: Subject Premature Ejaculation Profile (PEP) at Month 2
Description: Scores for perceived control over ejaculation, personal distress related to ejaculation, satisfaction with sexual intercourse and interpersonal difficulty related to ejaculation based on the subject PEP at month 2. Proportion of subjects with at least a 1 point category improvement in subject PEP domain scores from baseline to month 2.
Time Frame: 2 months
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
percentage of participants
  Control | 67.5 | 24.7
  Distress | 70.1 | 33.8
  Sexual satisfaction | 69.4 | 27.3
  Interpersonal difficulty | 75.8 | 42.9

9. Secondary Outcome: Subject Premature Ejaculation Profile (PEP) at Month 3
Description: Scores for perceived control over ejaculation, personal distress related to ejaculation, satisfaction with sexual intercourse and interpersonal difficulty related to ejaculation based on the subject PEP at month 3. Proportion of subjects with at least a 1 point category improvement in subject PEP domain scores from baseline to month 3.
Time Frame: 3 months
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
percentage of participants
  Control | 72.4 | 24.1
  Distress | 76.9 | 36.7
  Sexual satisfaction | 73.7 | 36.7
  Interpersonal difficulty | 77.6 | 59.5

10. Secondary Outcome: Partner Premature Ejaculation Profile (PEP) at Month 3
Description: Scores for perceived control over ejaculation, personal distress related to ejaculation, satisfaction with sexual intercourse and interpersonal difficulty related to ejaculation based on the partner PEP at month 3. Proportion of partners with at least a 1 point category improvement in partner PEP domain scores from baseline to month 3.
Time Frame: 3 months
Population: ITT
Measure: Number; unit: percentage of partners
Arm/Group | Double-Blind Active / Open-Label Active | Double-Blind Placebo / Open-Label Active
Number analyzed (Participants) | 167 | 82
percentage of partners
  Control | 68.9 | 40.8
  Distress | 64.9 | 50.0
  Sexual satisfaction | 62.8 | 32.9
  Interpersonal difficulty | 66.9 | 50.0

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events collected from randomisation to end of study
Description: Safety Population - all subjects that received the study drug.
Groups:
- Double-Blind Active: Double-blind Phase: Subjects will be randomised in a 2:1 ratio of PSD502 or placebo respectively if the patient meets all the entry criteria.
  PSD502, contains a mixture of lidocaine and prilocaine: PSD502 spray contains a mixture of lidocaine and prilocaine with Norflurane (HFA-134a) is used as both propellant and solvent. A single dose consists of 3 sprays applied to the glans penis.
  Approximately 5 minutes before intercourse the study spray (PSD502 or Placebo) can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
- Double-Blind Placebo: Double-blind Phase: Subjects will be randomised in a 2:1 ratio of PSD502 or placebo respectively if the patient meets all the entry criteria.
  PSD502 Placebo: The placebo is a metered dose aerosol spray that is identical in appearance to the PSD502 spray and contains the same propellant (norflurane) but has no lidocaine or prilocaine.
  Approximately 5 minutes before intercourse the study spray (PSD502 or Placebo) can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing.
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
- Open Label Phase: Subjects will all receive PSD502 if they wish to continue in the trial.
  PSD502, contains a mixture of lidocaine and prilocaine: PSD502 spray contains a mixture of lidocaine and prilocaine with Norflurane (HFA-134a) is used as both propellant and solvent. A single dose consists of 3 sprays applied to the glans penis.
  Approximately 5 minutes before intercourse the study spray (PSD502 or Placebo) can be applied and any excess should be wiped off with a damp cloth or tissue.
  During the initial 3 months double-blind phase of the study subjects should leave at least 24 hours between each dosing
  During the subsequent 5 months open label Phase of the study subjects may use the spray for up to a maximum of 3 sexual encounters (intercourse) in a 24 hour period. Each sexual encounter (intercourse) when the spray is used must be separated by at least 4 hour period.
Arm/Group | Double-Blind Active | Double-Blind Placebo | Open Label Phase
Serious Adverse Events (participants affected / at risk) | 1/167 | 1/82 | 4/223
Other Adverse Events (participants affected / at risk) | 9/167 | 0/82 | 8/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Active (N=167) | Double-Blind Placebo (N=82) | Open Label Phase (N=223)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease and myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
blood albumin, haematocrit, platelet count, protein total, RBC count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Active (N=167) | Double-Blind Placebo (N=82) | Open Label Phase (N=223)
Erectile dysfunction (Reproductive system and breast disorders) | 9 (14) | 0 (0) | 8 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and his/her results shall not be publicized or published in any form to cooperative publication without prior, written consent of Pharm-Olam or the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.